CLINICAL TRIAL: NCT00533572
Title: Recessive Dystrophic Epidermolysis Bullosa Screening for Possible Gene Transfer
Status: Terminated | Type: Observational
Why Stopped: Study was suspended until FDA approved the IND. Study has since been terminated and a new screening process has been implemented.
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Alfred Lane, Professor of Dermatology and of Pediatricsy, Emeritus, Stanford University
Other Study IDs: 97822; 8557
Record Dates: First submitted 2007-09-20; First posted 2007-09-21 (Estimated); Last update posted 2015-05-27 (Estimated); Status verified 2015-05

CONDITIONS: Epidermolysis Bullosa Dystrophica
MeSH Terms: conditions — Epidermolysis Bullosa Dystrophica

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional

SUMMARY:
Recessive Dystrophic Epidermolysis Bullosa (RDEB) is a severe inherited blistering skin disease caused by absence of type VII collagen. Patients with RDEB develop large, severly painful blisters and open wounds from minor trauma to their skin. In the future, we hope to start a gene transfer study on a specific group of RDEB subjects and we are screening subjects for that potential trial now.

DETAILED DESCRIPTION:
This study is a preparation for a gene transfer trial. In the gene transfer trial, we will transfect autologous RDEB keratinocytes with a type VII collagen containing retrovirus vector. We then plan to graft the genetically engineered and corrected autologous keratinocytes back on to wounds of the RDEB subject. We expect the grafts to attach as normal keratinocytes and replace the damaged skin with skin that is able to make type VII collagen and anchor normally to the dermis. We are trying to define the number of subjects 18 or older who meet the criteria for the gene transfer trial. We are offering the subjects the opportunity to be evaluated for the potential trial.

ELIGIBILITY:
Inclusion Criteria:1. Clinical diagnosis of RDEB by local dermatologist 2. 18 years of age or more and willing to give consent 3. Estimated to have at least 100 to 200 sq. cm. areas of open erosions on the trunk or extremities suitable for skin grafting 4. Ability to undergo adequate anesthesia to allow grafting procedures to take place 5. Parents are alive, do not have EB, and they are willing to give consent for genetic testing Exclusion Criteria:1. Medical instability limiting ability to travel to Stanford University Medical Center 2. Participation in another clinical trial without prior approval 3. The presence of medical illness expected to complicate participation and/or compromise the safety of this technique

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults with RDEB
Sampling Method: Non-Probability Sample
Enrollment: 1 (Actual)
Dates: Start 2007-08; Primary Completion 2008-08 (Actual); Study Completion 2008-08 (Actual)

PRIMARY OUTCOMES:
Disease documentation | 1 year
  Documentation of disease
documentation of disease | 1 year
  documentation of disease

CONTACTS AND LOCATIONS:
Overall Officials: Alfred T Lane, Principal Investigator — Stanford University
Locations (1):
- Stanford University School of Medicine, Stanford, California, United States